CLINICAL TRIAL: NCT05645302
Title: Intensive Monitoring Scheme of Lidocaine Cataplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Wei Xu, Principal Investigator, Qianfoshan Hospital
Other Study IDs: ZT-DBN-ZDJC-01
Record Dates: First submitted 2022-11-22; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Adverse Reaction to Drug
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients using Lidocaine Cataplasms
  Interventions: Drug: Lidocaine Cataplasms

INTERVENTIONS:
Drug: Lidocaine Cataplasms — The main ingredient of this product is lidocaine, the cream surface is white or almost white, the cream is evenly spread on the back, and the cream surface is covered with film.

SUMMARY:
In this center, retrospective research methods are used to collect data. Patients who had used Lidocaine Cataplasms at least once were included consecutively. Taking the time when the patient first used Lidocaine Cataplasms as the starting time (the study baseline), collect the demographic characteristics of the patient, the medication scheme of Lidocaine Cataplasms and other information, as well as the medication safety and other information from the first medication to the end of medication or discharge (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving Lidocaine Cataplasms from January 1, 2021 to April 1, 2022.

Exclusion Criteria:

* Unable to obtain complete medication information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have used Lidocaine Cataplasms at least 1 consecutive time between January 1, 2021 and April 1, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | January 1, 2021 - April 1, 2022
  Past medical history and other diseases that the researcher thinks have clinical significance. Collect the frequency, type, years, etc. of drinking and/or smoking, as well as the family history of diseases. Including white blood cell, red blood cell, hemoglobin, platelet count, etc. Including white blood cells, red blood cells, urine protein, urine sugar, etc. Including ALT, AST, ALP, TBil, GGT, BUN, Cr, etc. The researcher issued a prescription of lidocaine gel plaster according to the drug instructions, and recorded the indications, medication time, dose, frequency, drug batch number, etc. It includes all kinds of reactions unrelated to the treatment purpose during the study period, including symptoms, signs, laboratory abnormalities with clinical significance or special examinations.administration or discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China